CLINICAL TRIAL: NCT02611310
Title: Saudi Arabia - A Disease Registry Study to Prospectively Observe Treatment Patterns and Outcomes in Patients With HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study to Observe Treatment Patterns and Outcomes in Participants in Saudi Arabia With Human Epidermal Growth Factor Receptor 2 (HER2-Positive) Unresectable Locally Advanced or Metastatic Breast Cancer (LA/mBC)
Status: Terminated | Type: Observational
Why Stopped: Recruitment Target not met
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29618
Record Dates: First submitted 2015-11-19; First posted 2015-11-20 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with HER2-positive unresectable LA/mBC
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study.

SUMMARY:
This is a prospective, national, multicenter, non-interventional study designed to enroll participants who have an initial diagnosis of unresectable LA/mBC made up to 6 months prior to registry enrollment. These participants will be prospectively followed for at least 5 years after study enrollment to evaluate their anti-cancer treatments. Data on participants' previous anti-cancer treatments for breast cancer will be collected retrospectively at study entry.

ELIGIBILITY:
Inclusion Criteria:

* Initially diagnosed with HER2-positive unresectable LA/mBC no more than 6 months prior to enrollment
* Able to comply with the study protocol

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HER2-positive unresectable LA/mBC
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Up to 5 years
Overall Survival (OS) | Up to 5 years
Objective Response Rate (ORR) Per Anti-Cancer Treatment Regimen | Up to 5 years
Duration of Response (DoR) Per Anti-Cancer Treatment Regimen | Up to 5 years
Quality of Life, as Assessed by the EuroQol 5-Dimensions Questionnaire (EQ-5D) | Up to 5 years
Overall Health Status, as Assessed by the Functional Assessment of Cancer Therapy-Breast (FACT-B) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Saudi Arabia (3):
  - King Abdullah Medical City-Holy Makkah, Holy Makkah
  - National Guard King Abdulaziz Medical City; Oncology, Riyadh
  - King Fahad Medical City; Gastroentrology, Riyadh